CLINICAL TRIAL: NCT03045783
Title: Efficacy and Safety of Prophylactic Use of Antibiotics in Endoscopic Injection of Tissue Adhesive in Gastric Varices: A Multicenter Randomized Controlled Trial
Brief Title: Prophylactic Use of Antibiotics in Endoscopic Injection of Tissue Adhesive in Gastric Varices
Acronym: PUoA-EIoTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Lanzhou University Second Hospital (Other); Beijing Ditan Hospital (Other); Shandong Provincial Hospital (Other Government); Renmin Hospital of Wuhan University (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Shiyao Chen, Professor, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CSY-LCF2-2016
Record Dates: First submitted 2017-01-04; First posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Gastric Varices; Cirrhosis
Keywords: gastric varices; endoscopic injection of tissue adhesive
MeSH Terms: conditions — Esophageal and Gastric Varices; Fibrosis | interventions — Cefotiam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prophylactic use of antibiotics group (Experimental): Prophylactic use of antibiotics during endoscopic treatment, cefotiam 2.0g intravenous
  Interventions: Drug: Cefotiam
- On-demand group (No Intervention): Routine endoscopic examination and treatment. Antibiotics are not used during endoscopic treatment

INTERVENTIONS:
Drug: Cefotiam — Prophylactic use of antibiotics group：Prophylactic use of antibiotics during endoscopic treatment, cefotiam 2.0g intravenous
  Other Names: HaiTiShu
  Arms: Prophylactic use of antibiotics group

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of prophylactic use of antibiotics in endoscopic injection of tissue adhesive in gastric varices.

DETAILED DESCRIPTION:
Gastroesophageal variceal bleeding is the most common and life-threatening condition in patients with portal hypertension, which are susceptibility to bacterial infection. However, the prophylaxis use of antibiotics remained uncertain and lack of high level evidences.This study is a randomized controlled trial. The purpose of the study is to evaluate the efficacy and safety of prophylactic use of antibiotics in endoscopic injection of tissue adhesive in gastric varices.

ELIGIBILITY:
Inclusion Criteria:

* 18 y.o. ≤age≤75 y.o.;
* Diagnosis of esophageal gastric varices by gastroscopy;
* Cirrhotic gastroesophageal variceal bleeding underwent endoscopic injection of tissue adhesive;

Exclusion Criteria:

* age <18 y.o. or age > 75 y.o.;
* Never had the variceal bleeding episode before;
* Do not have endoscopic injection of tissue adhesive;
* The cefotiam contraindications: such as allergies, pregnancy etc;
* combined with other malignant tumor (not exclude patients with hepatocellular carcinoma who don't not need treatment at the moment);
* Known infection before endoscopic treatment (Fever, microbial cultures positive, et al.);
* Massive ascites or combined with other high risk factor that require prophylaxis use of antibiotics;
* Acute variceal bleeding within 5 days;
* Refuse to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 912 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-03 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
The incidence of infection after endoscopic treatment | 1 week
  Patients will receive body temperature, blood routine, inflammatory markers examination before and after endoscopic treatment

SECONDARY OUTCOMES:
Rebleeding rate | 2 months
  Patients will be followed up and receive an endoscopic examination after patients have been followed up for 2 months.
Mortality rate | 2 months
  The investigators observe the mortality events during 2 months
All clinical events | 2 months
  All clinical events were defined as occurrence rebreeding, ascitic fluid infection, portal vein thrombosis, or death.
Serum endotoxin | before and the first day after endoscopic treatment
inflammatory factors including IL-6, IL-8, TNF-a, IL-1beta，IL-2R, IL-10 | before and the first day after endoscopic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shiyao CHEN, M.D., Principal Investigator — Zhongshan Hospital, Fudan University, Shanghai
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No